CLINICAL TRIAL: NCT03636620
Title: Clinical Trial of Transcatheter Arterial Chemoembolization Combined With Radiofrequency/Microwave Ablation in Hepatocellular Carcinoma Beyond Milan Criterial
Brief Title: TACE Combined With RFA/MV Treatment in Hepatocellular Carcinoma Beyond Milan Criterial
Acronym: TACE+RFA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zheng-Gang Ren, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC-TACE+RFA/MV
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: TACE vs.TACE+RFA
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE group (Active Comparator): Transcatheter arterial chemoembolization
  Interventions: Device: Transcatheter arterial chemoembolization
- TACE+RFA/MV group (Experimental): Transcatheter arterial chemoembolization and radiofrequency /microwave ablation
  Interventions: Device: Transcatheter arterial chemoembolization; Device: radiofrequency ablation/microwave ablation

INTERVENTIONS:
Device: Transcatheter arterial chemoembolization — Transcatheter arterial chemoembolization
  Other Names: TACE
Device: radiofrequency ablation/microwave ablation — radiofrequency ablation/microwave ablation
  Other Names: RFA/MW
  Arms: TACE+RFA/MV group

SUMMARY:
This study was designed to evaluate the effectiveness of radiofrequency /microwave ablation in patients with hepatocellular carcinoma beyond Milan Criteria.

DETAILED DESCRIPTION:
The aim of this study is to included 120 patients with intermediate stage hepatocellular carcinoma beyond Milan criteria .These patients were randomizedly allocated to TACE treatment group or TACE+RFA/MV .The treatment effectiveness, local tumor control and survival outcome between the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* patients diganosed with hepatocellualr carcinoma beyond Milan criteria
* the presence of a single HCC tumor ≤7 cm in diameter, or multi-nodular HCC tumors (n ≤ 5) small than 7 cm in diameter;
* Child-Pugh A or B
* ECOG score 0-1;
* prothrombin time ≤16 s;
* white cell count ≥3,000/mm3, platelet count ≥40 x 109/L;Hb≥8.5 g/d; ALT/AST≤5×ULN;TB≤3mg/dl;alb≥2.8 g/dl ;Scr ≤2mg/dl

Exclusion Criteria:

* expected survival time < 12 months before random assignment;
* received anticancer surgery or procedure within one month before assignment;
* concomitant use of any other anticancer therapy(except immunotherapy and herbal medicine ) ;
* existence of portal of hepatic vein invation or extrahepatic metastases;existence of active infection ;
* upper gastrointestinal hemorrhage within one month ; .other serious illness or medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 46 months

SECONDARY OUTCOMES:
objective response rate | up to 46 months

CONTACTS AND LOCATIONS:
Overall Officials: zheng-gang Ren, doctor, Principal Investigator — Fudan University
Locations (1):
- liver cancer institute ,Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
no plan to make individual paticipant data available to other researchers